CLINICAL TRIAL: NCT05780619
Title: Diagnostic Performance of the Resistance Index (RI) for the Assessment of Cerebral Vasoreactivity in Transcranial Doppler
Acronym: REVACEIR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2022/SC-01
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stenosis; Occlusion
Keywords: Acetazolamide
MeSH Terms: conditions — Constriction, Pathologic; Bites and Stings | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with abnormal vasoreactivity
  Interventions: Diagnostic Test: Transcranial Doppler
- Patients with normal vasoreactivity
  Interventions: Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler — Measurement of resistance index on the middle cerebral artery (MCA) (index test) and the Holter (reference test). Patients will be randomized for order of tests

SUMMARY:
Routine revascularization of asymptomatic carotid stenosis is questionable as optimal medical therapy has significantly reduced the risk of stroke. Therefore, it is crucial to identify high-risk patients who may still benefit from carotid revascularization. In 2017, the ESC guidelines clarified the criteria associated with a high risk of stroke despite optimal treatment to consider a revascularization procedure, including altered cerebral vasoreactivity. However, cerebral vasoreactivity using transcranial Doppler ultrasound is reserved for qualified centers. It requires a technical platform and trained personnel, is time-consuming and generally not readily available.

A simpler test is therefore necessary. The goal is to quickly and easily detect patients with normal vasoreactivity who do not benefit from the cerebral vasoreactivity test (reference standard) and to reserve the time-consuming cerebral vasoreactivity test for patients likely to have altered vasoreactivity.

The hypothesis of the study is that on a routine measure in transcranial echo-Doppler, the resistance index (RI), can predict the response to the cerebral vasoreactivity test. With this new test, it will be possible to select patients who do not benefit from pharmacological cerebral vasoreactivity testing ("true negatives"). Thus, the time-consuming cerebral vasoreactivity test will be reserved only for patients with a possibility of impaired vasoreactivity.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Stenosis ≥ 70% in diameter reduction in NASCET equivalent or occlusion of atheromatous origin of the cervical internal carotid artery, asymptomatic or symptomatic.
* Presence of a temporal window sufficient to record the homolateral and contralateral middle cerebral artery.
* Patient of legal age with free and informed consent.
* Patient who has signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Contraindication to Acetazolamide Diamox® injection.
* Absence of temporal acoustic window (non visualization of the cerebral parenchyma, no recordable intracranial vessel).
* Insufficient temporal window (visualizable brain parenchyma, no recordable MCA)
* Internal or common carotid artery stenosis ≥70% or occlusion, contralateral to the primary lesion.
* Stenosis ≥50% of the middle cerebral artery homolateral or contralateral to the cervical lesion.
* Patient in exclusion period determined by another study.
* Patient under court protection, guardianship, or conservatorship.
* Patient refusing to sign the consent form.
* Patient unable to express his or her will (dementia, disturbed consciousness, etc.)
* Patient for whom it is impossible to give informed information for health reasons or because of a language barrier.
* Pregnant, parturient, or breastfeeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out at the University Hospital of Nîmes in the department of explorations and vascular medicine (EMV), for patients referred for HRV measurement with a significant stenosis or occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Specificity of the difference in average resistance index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Sensitivity of the difference in average resistance index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Positive predictive value of the difference in average resistance index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Negative predictive value of the difference in average resistance index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test

SECONDARY OUTCOMES:
Sensitivity of the difference in average Gosling's pulsatility index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Specificity of the difference in average Gosling's pulsatility index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Positive predictive value of the difference in average Gosling's pulsatility index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Negative predictive value of the difference in average Gosling's pulsatility index (delta) between the middle cerebral artery (MCA) on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity | Day 1
  normal vasoreactivity defined as an increase in the mean of the maximum velocities > 30% measured by the cerebral vasoreactivity reference test
Correlation between delta resistance index and percentage response of vasoreactivity reference test | Day 1
  correlation coefficient
Correlation between delta Gosling's pulsatility index and percentage response of vasoreactivity reference test correlation coefficient | Day 1
  correlation coefficient
Sensitivity of the difference in average Gosling's pulsatility index (delta) between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Specificity of the difference in average Gosling's pulsatility index (delta) between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Positive predictive value oof the difference in average Gosling's pulsatility index (delta) between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Negative predictive value of the difference in average Gosling's pulsatility index (delta) between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Sensitivity of the difference in average resistance index between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Specificity of the difference in average resistance index between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Positive predictive value of the difference in average resistance index between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1
Negative predictive value of the difference in average resistance index between the MCA on the M1 segment contralateral and homolateral to the carotid lesion, to detect normal vasoreactivity in symptomatic versus asymptomatic stenosis | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Coudray, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No